CLINICAL TRIAL: NCT05086861
Title: Oesophageal Pacing to Check Left Atrial Posterior Wall Isolation: A Pilot Study
Brief Title: Oesophageal Pacing to Check Left Atrial Posterior Wall Isolation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15/P/094
Record Dates: First submitted 2019-08-29; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2020-12

CONDITIONS: Persistent Atrial Fibrillation; Atrial Fibrillation Ablation
Keywords: Oesophageal Pacing; Hybrid Ablation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oesophageal Pacing Arm (Experimental): Patients undergoing atrial fibrillation ablation to isolate the left atrial posterior wall via catheter or staged hybrid ablation.
  Interventions: Device: Oesophageal pacing after left atrial posterior wall isolation

INTERVENTIONS:
Device: Oesophageal pacing after left atrial posterior wall isolation — Following AF ablation with the aim of isolating the left atrial posterior wall oesophageal pacing and sensing is performed to check for left atrial posterior wall. entrance and exit block.

SUMMARY:
Patients undergoing hybrid AF ablation second stage catheter ablation have the posterior left atrium mapped to see it if is electrically isolated. This is done via a standard electrophysiogical study in accordance with routine clinical practice.

Investigators propose to check left atrium posterior wall isolation via oesophageal pacing and compare this to findings from invasive study

DETAILED DESCRIPTION:
Oesophageal temporary pacing of the heart is an established treatment in heart block and several catheters are licenced for this purpose with minimal procedural risks. Due to the position of the oesophagus, pacing from the oesophagus could sense and pace the posterior left atrium. If the posterior wall could be demonstrated to be electrically isolated with oesophageal pacing then invasive electrophysiological study such as the second stage of a hybrid AF ablation would be unnecessary.

This would save patients from undergoing invasive left atrial mapping and exposure to the consequent risks of the procedure.

ELIGIBILITY:
Inclusion Criteria: • subjects capable of giving informed consent,

* Male or female
* Aged between 18 and 80 years
* Undergoing ablation under general anaesthetic with planned isolation of the left atrial posterior wall or who have previously undergone either catheter or surgical ablation for AF with LA posterior wall isolation

Exclusion Criteria:

* Unable or willing to give fully informed written consent
* Turned down for general anaesthetic
* Pregnancy
* Terminal illness
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Left atrial posterior wall isolation | Through study completion, an average of 4 years
  Measured via invasive left atrial mapping

SECONDARY OUTCOMES:
Complication rate | Through study completion, an average of 4 years
  Documentation of the number of complications caused by the oesophageal pacing procedure
Feasibility of using device | Through study completion, an average of 4 years
  The success rate of left atrial posterior wall isolation.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Haywood, MD, Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Derriford Hospital, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No